CLINICAL TRIAL: NCT07166328
Title: RELATIONSHIP BETWEEN AXIAL AND FRONTAL BACK ASYMMETRY WITH SELF BODY IMAGE IN ADOLESCENT IDIOPATHIC SCOLIOSIS
Brief Title: Frontal/Axial and Self Body Image In Scoliosis
Status: Recruiting | Type: Observational
Sponsor: Al Hayah University In Cairo (Other)
Responsible Party: Principal Investigator, Sara Adel Abdelrahman Zaki, Demonstrator of Physical Therapy, Al Hayah University In Cairo
Other Study IDs: Fro-axial2024
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Scoliosis Idiopathic Adolescent; Scolosis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- One group - adolescent idiopathic scoliosis: Measure frontal and axial back asymmetry by BACKSCNR with self body image by TAPS questionnaire
  Interventions: Device: BACKSCNR , measure the deviations of frontal and axial back asymmetry in AIS

INTERVENTIONS:
Device: BACKSCNR , measure the deviations of frontal and axial back asymmetry in AIS — BACKSCNR is a non-invasive surface topography device designed to assess spinal deformities, particularly scoliosis. It uses optical scanning technology to capture the three-dimensional shape of the back without radiation exposure.

SUMMARY:
What is the relationship between frontal and axial back asymmetric parameters with self body image in adolescent idiopathic scoliosis Age This study will investigate the relationship between frontal and axial back asymmetry with self body image in adolescent idiopathic scoliosis Delimitations : patients will be diagnosed by orthopedic surgeon with adolescent idiopathic scoliosis Delimitations Age 11 to 18 years BMI fron 20 to 24.9kg/m2 Moderate cobbs angle 25-45 degrees Major thoacic curve Self body image will be ass by TAPS questionnaire which evaluate self image and satisfaction

ELIGIBILITY:
Inclusion Criteria:

* Both gender's adolescent idiopathic scoliosis Age from 11 to 18 years Body mass index 20-25Kg/m2 Moderate cobb's angle 25/45 degree Participation should be normal ambulatory Major thoracic curve

Exclusion Criteria:

* leg length discrepancy Any mental condition Defects of spinal vertebrae Previous history of spine or lower extremities surgery

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescent idiopathic scoliosis , age 11 to 18 years , cobb more than 10 degrees-no congenital or neuromuscular disorders.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Frontal plane back asymmetry | At baseline
  Frontal plane back asymmetry will be measured using BACKSCNR. The device quantifies deviations of the trunk in the frontal plane. Higher values indicate greater asymmetry.
Axial trunk deviations | At baseline
  Axial trunk deviations will be measured using BACKSCNR. The device quantifies rotational deviations of the trunk in the transverse plane. Higher values indicate greater asymmetry.
Self-perceived body image (TAPS questionnaire) | At baseline
  Self-body image will be assessed using the Trunk Appearance Perception Scale (TAPS), a validated questionnaire for individuals with scoliosis. The TAPS measures the patient's subjective perception of trunk deformity in different views. Scores range from 1 to 5, with lower scores indicating a perception of greater deformity and higher scores indicating a perception closer to normal trunk appearance.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy Alhayah university, New Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No